CLINICAL TRIAL: NCT01606592
Title: Phase 2/3 Study of Panic Control Treatment vs Panic-Focussed Psychodynamic Psychotherapy Under Randomized and Self-Selection Conditions
Brief Title: Psychotherapy Outcome and Self-selection Effects in Panic Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: POSE
Record Dates: First submitted 2012-03-19; First posted 2012-05-25 (Estimated); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Panic Disorder (With or Without Agoraphobia)
MeSH Terms: conditions — Panic Disorder | interventions — Waiting Lists

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Randomized Panic Control Treatment (Experimental): Patients who have been randomized to the randomization condition are assigned to PCT
  Interventions: Behavioral: Panic Control Treatment (PCT)
- Randomized Panic-Focused Psychodynamic Psychotherapy (Experimental): Patients who have been randomized to the randomization condition are assigned to PFPP
  Interventions: Behavioral: Panic-Focused Psychodynamic Psychotherapy (PFPP)
- Self-selected Panic Control Treatment (Experimental): Patients who have been randomized to the self-selection condition choose PCT
  Interventions: Behavioral: Panic Control Treatment (PCT)
- Self-selected Panic-Focussed Psychodynamic Psychotherapy (Experimental): Patients who have been randomized to the self-selection condition choose PFPP
  Interventions: Behavioral: Panic-Focused Psychodynamic Psychotherapy (PFPP)
- Waiting-list (Experimental): Patients who have been randomized to the waiting-list are offered sparse contact over telephone for 12 weeks and are then re-randomized to one of the other four arms
  Interventions: Other: Waiting-list

INTERVENTIONS:
Behavioral: Panic Control Treatment (PCT) — Manualized, 13 sessions (60 min, sometimes extended to 90-120) completed in 12-16 weeks. Total duration 840-1080 min.
  Arms: Randomized Panic Control Treatment; Self-selected Panic Control Treatment
Behavioral: Panic-Focused Psychodynamic Psychotherapy (PFPP) — Manualized, 19-24 sessions (45 min) completed in 12-16 weeks. Total duration 855-1080 min.
  Arms: Randomized Panic-Focused Psychodynamic Psychotherapy; Self-selected Panic-Focussed Psychodynamic Psychotherapy
Other: Waiting-list — Sparse telephone contact during 12 weeks, then re-randomization
  Arms: Waiting-list

SUMMARY:
The efficacy of two forms of psychotherapy with panic disordered patients, a cognitive-behavioral and a psychodynamic one, are compared under two different, randomized conditions: randomization or self-selection. The basic hypotheses are that the efficacy of both treatments is higher and that the efficacy difference is smaller under self-selection than randomized conditions.

DETAILED DESCRIPTION:
After thorough assessment persons with a panic disorder diagnosis are randomly assigned to three arms: one randomization, one self-selection, and one a low-contact waiting list one. In the randomization arm (R) 95 persons are randomly assigned to Panic Control Treatment (PCT) or Panic-Focused Psychodynamic Psychotherapy (PFPP); in the self-selection arm (SS) 95 persons are offered, after adequate information, to choose which of the two they prefer. Twenty-six persons are initially randomized to a three-month waiting list (with sparse contact over telephone), after which they will be re-randomized, either to further randomization (to PCT or PFPP) or to self-selection. The four groups (R/PCT; R/PFPP; SS/PCT; SS/PFPP) will be compared on the basis of intake and repeated outcome/follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

* A Diagnostic and Statistical Manual (DSM-V) diagnosis of Panic Disorder, with or without Agoraphobia
* Age between 18 and 60
* Willingness to stop other on-going psychotherapy treatments and to refrain from nonstudy treatments during follow up
* Ability to complete the active treatment phase (not including follow-ups) within 16 weeks

Exclusion Criteria:

* Active substance dependence (6 months remission necessary)
* Current psychosis, delusions, mania, or active addiction
* Acute suicidality
* A history and clinical presentation of at least one clinically-significant medical condition if, due to their cognitive or physical impairments, they are unable to fully participate in the psychotherapy treatments being offered
* Active involvement in a legal dispute related to their mental health issues
* Three or more unexcused absences

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 216 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2021-02 (Actual)

PRIMARY OUTCOMES:
Change on Panic Disorder Severity Scale (PDSS; Shear et al., 1997) | Growth curve analysis across intake and follow up at termination and 6, 12 and 24 months after termination
Change in occupational status | Growth curve analysis across intake and follow up at termination and 6, 12 and 24 months after termination
Change in absence from work due to sickness | Growth curve analysis across 3 months before intake, intake and follow up at termination and 6, 12 and 24 months after termination

SECONDARY OUTCOMES:
Change on Mobility Inventory for Agoraphobia (MI, Chambless et al, 1985) | Growth curve analysis across intake and follow up at termination and 6, 12 and 24 months after termination
Change in health care utilization (number of medical contacts, and emergency visits, medication) | Growth curve analysis across 3 months before intake, intake and follow up at termination and 6, 12 and 24 months after termination
Change on Clinical Outcomes in Routine Evaluation Scale(CORE; Evans et al., 2000) | Growth curve analysis across intake and follow up at termination and 6, 12 and 24 months after termination
Change on Montgomery Asberg Depression Rating Scale (MADRS-S; Montgomery & Asberg, 1979) | Growth curve analysis across intake and follow up at termination and 6, 12 and 24 months after termination

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Sandell, PhD, Principal Investigator — Lund University
Locations (1):
- Lund University, Lund, Sweden

REFERENCES:
- [Derived] Nilsson T, Falkenstrom F, Perrin S, Svensson M, Johansson H, Sandell R. Exploring termination setback in a psychodynamic therapy for panic disorder. J Consult Clin Psychol. 2021 Sep;89(9):762-772. doi: 10.1037/ccp0000678. PMID 34591549
- [Derived] Svensson M, Nilsson T, Perrin S, Johansson H, Viborg G, Sandell R. Preferences for panic control treatment and panic focused psychodynamic psychotherapy for panic disorder - who chooses which and why? Psychother Res. 2021 Jun;31(5):644-655. doi: 10.1080/10503307.2020.1839686. Epub 2020 Nov 5. PMID 33148129
- [Derived] Svensson M, Nilsson T, Johansson H, Viborg G, Perrin S, Sandell R. Psychometric analysis of the Swedish panic disorder severity scale and its self-report version. Nord J Psychiatry. 2019 Jan;73(1):58-63. doi: 10.1080/08039488.2018.1554699. Epub 2019 Jan 14. PMID 30636466
- [Derived] Sandell R, Svensson M, Nilsson T, Johansson H, Viborg G, Perrin S. The POSE study - panic control treatment versus panic-focused psychodynamic psychotherapy under randomized and self-selection conditions: study protocol for a randomized controlled trial. Trials. 2015 Mar 31;16:130. doi: 10.1186/s13063-015-0656-7. PMID 25873067